CLINICAL TRIAL: NCT01376466
Title: The Impact Of Computed Tomography On The Diagnoses Of Acute Appendicitis
Brief Title: Impact of CT on Diagnosis of Acute Appendicitis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Herning Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M-20080129
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Acute Appendicitis
Keywords: acute appendicitis; diagnosis; computed tomography
MeSH Terms: conditions — Appendicitis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with acute appendicitis: Patients who have been clinically diagnosed to have acute appendicitis
  Interventions: Other: CT scanning

INTERVENTIONS:
Other: CT scanning — CT image of the abdomen included the area between the 3rd. lumber vertebra and the top of acetabulum. A liter of contrast mixed with normal salin will be given by rectal catheter 20 minutes before CT image is taken.
  Other Names: CT scanning of the abdomen

SUMMARY:
The purpose of this study is to determine whether computed tomography is reliable investigation in the diagnosis of acute appendicitis.

DETAILED DESCRIPTION:
The aim of this study is to

1. evaluate CT scan validity for the diagnosis of acute appendicitis.
2. compare the difference in evaluation of CT-scan result between radiologist on call and consultant radiologist with CT experience.
3. illustrate difficulties associated with practical implementation of CT-scan in relation to other activities in radiology department and O.R. (logical & organizational).
4. illustrate patients experiences about the study (pain, discomfort & other information

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been admitted and diagnosed as having acute appendicitis

Exclusion Criteria:

* Patients under the age of 18 years.
* Pregnancy.
* Uncooperative patients (senile dementia, mentally ill).
* Not speaking Danish.
* Does not wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients with acute appendicitis.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens R Madsen, MD, Study Director — Consultant surgeon
Locations (1):
- Herning Hospital, Herning, Herning, Denmark